CLINICAL TRIAL: NCT07045233
Title: A Clinical Study on the Use of the Sentinel Cerebral Protection Device During TAVR for the Prevention of Procedure-Related Stroke
Acronym: SENTINEL-TAVR
Status: Enrolling by invitation | Type: Observational
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2024-KJCX04-04
Record Dates: First submitted 2025-06-22; First posted 2025-07-01 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2024-08

CONDITIONS: Stroke; Transcatheter Aortic Valve Replacement (TAVR); Aortic Stenosis Treated With TAVI
Keywords: stroke; Cerebral Protection Device; TAVR
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Sentinel® Cerebral Protection System — Deploy a Sentinel cerebral protection device during TAVR for patient with aortic stenosis.
Diagnostic Test: MRI — Patients receive head MRI before and after the surgery in order to determine the stroke incidence.

SUMMARY:
After more than a decade of development, transcatheter aortic valve replacement (TAVR) is now a standard, guideline-recommended treatment for all symptomatic patients with severe aortic stenosis, regardless of their surgical risk. However, stroke remains a risk for these patients after TAVR. Given its severe impact-significantly increasing post-procedure mortality and severely affecting quality of life-preventing TAVR-related stroke is an urgent problem we need to solve.

The Sentinel Cerebral Protection Device is a percutaneous dual-filter brain protection system. During the procedure, the Sentinel device's filters capture blood clots and tissue debris. After the operation, the captured clots and debris are removed from the body along with the device. Its safety and effectiveness have been validated. Therefore, this project plans to conduct a multi-center registry clinical study to:

Develop a widespread neurological risk prediction model. Create a strict, standardized prevention protocol. Boost awareness of perioperative stroke prevention during TAVR. Provide practical clinical experience. By doing so, we aim to better prevent strokes in patients undergoing TAVR.

ELIGIBILITY:
Inclusion Criteria:

* Patients who meet the surgical indications for Transcatheter Aortic Valve Replacement (TAVR), diagnosed as symptomatic severe aortic stenosis, receive a Sentinel Cerebral Protection System during the procedure, and are adult patients who have been informed and consented to participate in this study.

Exclusion Criteria:

* History of cerebral disease within 1 year prior to the procedure (e.g., stroke, cerebral hemorrhage, brain tumor, encephalitis, traumatic brain injury, or other craniocerebral-related diseases).

History of previous open-chest surgery or previous heart valve replacement. Patients with left ventricular ejection fraction ≤ 30%. Presence of contraindications for MRI examination. Patients with claustrophobia. Patients unable to comply with follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in China
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
The Rate of Stroke Through 72 Hours Post TAVR Procedure or Discharge (Whichever Comes First) | From enrollment to 72 hours post surgery or discharge (whichever comes first)
  All stroke (hemorrhagic, ischemic, or undetermined status; disabling or nondisabling) through 72 hours post TAVR procedure or discharge (whichever comes first), as adjudicated by an independent Clinical Events Committee (CEC) and using Neurologic Academic Research Consortium (NeuroARC) definitions.

CONTACTS AND LOCATIONS:
Overall Officials: Yongquan Xie, Principal Investigator — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (1):
- Fuwai Hospital, Beijing, China